CLINICAL TRIAL: NCT06737341
Title: Effect of Bupivacaine Liposomes or Bupivacaine for Ultrasound-guided CMB on Postoperative Analgesia in Laparoscopic Hepatobiliary Pancreatic Surgery: a Prospective, Single Blind, Completely Randomized, Active Controlled Clinical Trial
Brief Title: Bupivacaine Liposomes or Bupivacaine for CMB on Postoperative Analgesia in Laparoscopic Hepatobiliary Pancreatic Surgery
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Wei Mei, MD,Department of Anesthesiology, Tongji Hospital, Tongji Medical College, HUST, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Tongji Hospital 20241030
Record Dates: First submitted 2024-12-09; First posted 2024-12-17 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Bupivacaine; Ultrasound-Guided; Analgesia, Postoperative; Opioids
Keywords: Bupivacaine Liposome; Costal Margin Block; Laparoscopic Hepatobiliary Pancreatic Surgery
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- bupivacaine liposomes(BL) (Experimental): 20ml of bupivacaine liposomes + 10ml 0.75% bupivacaine hydrochloride + 20ml normal saline for ultrasound-guided bilateral costal margin block. Block method: First, the high-frequency ultrasound probe is placed in the direction of the parasternal line parallel to the costal edge, and find the image of the costal cartilage and rectus abdominis space 。The needle was inserted along the medial side of the rectus to the lateral plane, and 15 ml of local anesthetic was injected between the costal cartilage and rectus abdominis space 。The ultrasound probe was then moved along the costal margin to the axillary front, flush with the tenth rib, and 10 ml of local anesthetic was injected in the plane between the tenth rib and the extraabdominal oblique muscle 。Similarly, perform ultrasound-guide costal rim block on the other side.
  Interventions: Drug: Bupivacaine Liposomes(BL)
- bupivacaine(B) (Active Comparator): 10 ml of 0.75% bupivacaine hydrochloride + 40ml normal saline for ultrasound-guided bilateral costal margin block in the same method as the experimental group
  Interventions: Drug: Bupivacaine(B)

INTERVENTIONS:
Drug: Bupivacaine Liposomes(BL) — 20ml of bupivacaine liposomes (266mg) + 10 ml of bupivacaine 0.75% hydrochloride + 20ml saline for ultrasound guided CMB.
  Arms: bupivacaine liposomes(BL)
Drug: Bupivacaine(B) — 10 ml of 0.75% bupivacaine hydrochloride + 40ml normal saline for ultrasound-guided bilateral costal margin block
  Arms: bupivacaine(B)

SUMMARY:
Numerous studies have confirmed that regional analgesia using peripheral nerve block has great potential for perioperative analgesia in abdominal surgery. Ultrasound guided costal margin block (CMB) is a new regional anesthesia technique that has been proven to compensate for the analgesic effects of regional analgesia techniques such as transverse abdominal muscle plane (TAP) and rectus abdominis sheath (RSB) on mid abdominal incisions, but it is difficult to meet the analgesic needs of anterior and outer abdominal wall incisions. According to relevant anatomy and research, the application of local anesthetics along the rib margin under the rectus abdominis muscle or under the external oblique muscle on the rib surface can block the lateral and anterior cutaneous branches of the thoracoabdominal nerve, known as CMB. Ultrasound guided CMB requires the injection of local anesthetics onto the surface of the rib along the plane below the rectus abdominis and oblique muscles, covering most of the upper abdominal incision pain. However, there are few reports on other types of upper abdominal surgeries such as liver, gallbladder, and pancreas surgeries.

Bupivacaine liposomes are an important innovation, which encapsulate bupivacaine in polycystic liposomes using DepoFoam technology to achieve slow drug release and effectively prolong pain relief time by up to 72 hours. This ultra long acting local anesthetic has significant advantages in reducing opioid use, improving analgesic satisfaction, reducing complications, and shortening hospital stays, and has been applied in the ERAS concept.

The investigators designed a prospective, single blind, randomized, active controlled clinical trial to investigate the effect of bupivacaine liposomes in combination with bupivacaine mixture or bupivacaine alone for ultrasound-guided bilateral CMB on postoperative analgesia in patients undergoing laparoscopic hepatobiliary pancreatic surgery. Our main hypothesis is that the use of bupivacaine liposomes and a mixture of bupivacaine for ultrasound-guided CMB in a multimodal analgesia regimen can more effectively reduce the dosage of intravenous patient-controlled analgesia (PCA) opiates within 72 hours after laparoscopic hepatobiliary pancreatic surgery compared to using bupivacaine alone. Secondary outcomes include the dosage of PCA opiates within 24-48 hours, pain score values, patient satisfaction, adverse reactions, and complications.

DETAILED DESCRIPTION:
All participators were randomized into two groups using a complete randomization allocation method: the trial group and the control group. An investigator introduced the study to the study before surgery and informed consent was obtained. The investigators educate patients on how to use the VAS scale to express pain intensity and instruct patients on how to use the postoperative analgesia pump. General anesthesia with endotracheal intubation or laryngeal mask before the nerve block. Standard analgesic protocol: sufentanil (0.5 μg/ kg) + remifentanil (0.1-0.2 μg / kg/min) + flurbiprofen ester (50mg); intravenous analgesia pump (PCIA) or analgesic with opioids and non-steroidal anti-inflammatory drugs as needed. All patients underwent ultrasound-guided bilateral costal margin block (CMB). Test group: 20ml bupivacaine liposomes +10ml 0.75% bupivacaine hydrochloride + 20ml normal saline, for ultrasound-guided CMB. Control group: 10 ml of 0.75% bupivacaine hydrochloride + 40ml of normal saline, with ultrasound-guided CMB.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old ASA Level I-III Laparoscopic Hepatobiliary Pancreatic Surgery

Exclusion Criteria:

* Body Mass Index (BMI) ≥ 30 kg/m ² or ≤ 15 kg/m ² Known alcohol or drug abuse History of upper abdominal surgery Congenital coagulation dysfunction Localized or systemic infection Peripheral neuropathy Unable to understand the research plan

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-08 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Overall Opioid Consumption | up to 3 days
  Main outcome measure: Postoperative 72 hour intravenous patient-controlled analgesia opioid dosage.

SECONDARY OUTCOMES:
Pain intensity | up to 3 days
  Pain intensity will be assessed using the Numerical Rating Scale (NRS), a 0-10 scale where 0 represents no pain and 10 represents the worst imaginable pain. Pain intensity will be measured during rest (supine position) and activity (shifting from supine position to lateral position) at 5 time points: at Post Anesthesia Care Unit(PACU), 6 hours, 24 hours, 48 hours，and 72 hours post-surgery
Cumulative use of opioid drugs | up to 2 days
  Cumulative use of opioid drugs for 24-48 hour intravenous patient-controlled analgesia
Other indicators | through study completion, an average of 10 day
  The incidence of postoperative pulmonary complications (including pneumonia, hypoxemia, and atelectasis), postoperative sleep quality (Pittsburgh Sleep Quality Scale), patient satisfaction with postoperative analgesic treatment (0-10 scale, 0 for very dissatisfied, 10 for very satisfied), time of first ambulation after surgery, time of first anal exhaust after surgery, length of hospital stay, and adverse events such as opioid related dizziness, nausea, and vomiting, as well as block related complications.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Mei, MD, Principal Investigator — Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Department of Anesthesiology, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology. 1095 Jiefang Avenue, Wuhan City, Hubei Province, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes
individual participant data sets to be shared will include all collected individual participant data that underlie the results reported in any publications resulting from the trial. This would typically include data related to pain relief, opioid analgesic consumption, incidence of complications, and any other relevant outcomes assessed at multiple time points within 72 hours after surgery.
Supporting Information: Study Protocol
Time Frame: From February 1,2025 to February 1,2027
Access Criteria: The IPD and any additional supporting information will be shared with qualified researchers upon request. Access will be granted for the purpose of conducting further analyses related to the outcomes of the clinical trial, such as but not limited to, pain relief, opioid analgesic consumption, and complications. Requests for access will be reviewed by the principal investigators and designated research personnel to ensure that the proposed analyses align with the objectives of the study and maintain participant confidentiality. Access to the data will be provided through a secure mechanism that safeguards the privacy and integrity of the individual participant data.